CLINICAL TRIAL: NCT01833195
Title: Outcomes AlloMap Registry Study: the Clinical Long-term Management and Outcomes of Heart Transplant Recipients With Regular Rejection Surveillance Including Use of AlloMap Gene-expression Profiling Testing
Brief Title: Outcomes AlloMap Registry: the Long-term Management and Outcomes of Heart Transplant Recipients With AlloMap Testing
Acronym: OAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00003
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Transplant Failure; Cardiac Transplant Rejection; Heart Diseases
Keywords: molecular diagnostics; heart transplantation; risk factors; prognosis
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — RNA isolated from peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart transplant recipients: Heart transplant rejection surveillance including AlloMap testing

SUMMARY:
The objective of this registry is to observe short and long term clinical outcomes in heart transplant recipients who receive regular AlloMap testing as part of allograft rejection surveillance.

DETAILED DESCRIPTION:
The standard of care in adult heart transplant recipients has been to perform periodic endomyocardial biopsies for surveillance for rejection. Because of the risks and discomforts associated with the biopsy procedure, a non-invasive test (AlloMap) based on gene-expression profiling of peripheral blood was developed and introduced in 2005 to identify heart transplant recipients who have a low probability of rejection at the time of protocol surveillance testing. The schedule of AlloMap surveillance testing has been derived from the customary timing of surveillance biopsies: e.g. at 1 to 2 month intervals for patients who are 6 and 12 post-transplantation, and at 3, 4 or 6 months after the first year post-transplantation.

In the large multicenter IMAGE (Invasive Monitoring Attenuation by Gene Expression Profiling) 602 patients in the United States who had undergone cardiac transplantation at least 6 months prior were randomized 1:1 to either surveillance with routine biopsy or AlloMap testing. Patients in both groups were also monitored with echocardiography. A primary outcome event was defined as an episode of rejection with hemodynamic compromise, graft dysfunction due to other causes, death or retransplantation. Over a median follow-up period of 19 months, 297 patients who were monitored with AlloMap and 305 patients who underwent routine biopsies had similar 2-year cumulative rates of events (14.5% and 15.3%, respectively; hazard ratio with gene-expression profiling, 1.04; 95% confidence interval, 0.67 to 1.68).

This Outcomes AlloMap Registry (OAR) study is designed to collect similar clinical outcomes information as studied in IMAGE, in a larger cohort of patients (approximately 2000) followed for up to 5 years. At each routine clinic visit, key clinical features such as rejection surveillance management schedules, testing results (e.g. blood levels of immunosuppressive agents), and AlloMap scores will be collected. This larger and longer term follow-up dataset is intended to enable further elucidation, through analyses techniques such as multivariate Cox proportional hazards models, of the surveillance management features which may be associated or contribute to the most favorable long term outcomes of the heart recipients.

ELIGIBILITY:
Inclusion Criteria:

* New and existing heart transplant recipients ≥ 2 months (≥ 55 days) post-transplant receiving post-transplant care at the enrolling centers for interim surveillance monitoring that includes AlloMap testing

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Heart transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 2444 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Vital status of heart transplant recipient | 5 Years
  Hospitalizations and causes (i.e. infections or graft dysfunction (classified as: acute cellular rejection, antibody mediated rejection , cardiac allograft vasculopathy or non specific etiology of graft dysfunction
  Cancers (newly diagnosed and/or recurrent): onset and classification of types of cancers

SECONDARY OUTCOMES:
Surveillance visit schedules and patient management parameters | 5 Years
  Endomyocardial biopsy and histology grades of rejection; left ventricular echocardiograms and ejection fractions; maintenance immunosuppressive drugs categories and doses/ blood levels; AlloMap scores and score patterns

CONTACTS AND LOCATIONS:
Overall Officials: James P Yee, MD, PhD, Study Director — CareDx, Inc., Brisbane, CA
Locations (36):
- United States (36):
  - Mayo Clinic, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Florida,, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mid America Heart Institute - St. Luke's Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor St. Lukes, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Intermountain Heart Institute, Murray, Utah
  - Inova Heart & Vascular Institute, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Shah MR, Starling RC, Schwartz Longacre L, Mehra MR; Working Group Participants. Heart transplantation research in the next decade--a goal to achieving evidence-based outcomes: National Heart, Lung, And Blood Institute Working Group. J Am Coll Cardiol. 2012 Apr 3;59(14):1263-9. doi: 10.1016/j.jacc.2011.11.050. PMID 22464255
- [Background] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- [Result] Kanwar, M. et al: Correlation of Longitudinal Gene-Expression Profiling Score to Cytomegalovirus (CMV) Infection: Results from the Outcomes AlloMap Registry (OAR). ISHLT 35th Annual Meeting and Scientific Sessions. 2015 April 13-18, 2015; Nice, France. *2015 American Transplant Congress. May 2-6, 2015; Philadelphia, PA. Poster.
- [Result] Teuteberg, J. et al; Gene-Expression Profiling to Monitor for Rejection-Which Patients are Being Offered This Strategy? ISHLT 35th Annual Meeting and Scientific Sessions. 2015 April 13-18, 2015; Nice, France. 2015. *American Transplant Congress. May 2-6, 2015; Philadelphia, PA. Poster.
- [Result] Sulemanjee, N. et al; Gender-Mismatched Heart Transplants and Gene Expression Profiling Score-Lessons Learned from the Outcomes AlloMap Registry (OAR). ISHLT 35th Annual Meeting and Scientific Sessions. 2015 April 13-18, 2015; Nice, France. 2015 *American Transplant Congress. May 2-6, 2015; Philadelphia, PA. Poster.
- [Result] Kanwar, M. et al; Impact of Cytomegalovirus Infection on Longitudinal Gene-Expression Profiling Score: Results from the Outcomes AlloMap Registry. 2016 ISHLT 36th Annual Meeting and Scientific Sessions. April 27-30, 2016; Washington, DC.
- [Result] Teuteberg, JJ. et al; Higher Rate of Hospitalizations for Infection and Cancer Then Rejection in Low Risk Heart Transplant Patients Followed by Gene Expression Profiling. 2016 ISHLT 36th Annual Meeting and Scientific Sessions. April 27-30, 2016; Washington, DC.
- [Result] Teuteberg, JJ. et al; Gene Expression Profiling Score and the Risk of Infection in Heart Transplant. 2016 American Transplant Congress. June 12, 2016; Boston, MA Poster
- [Result] Teuteberg, J., Shullo, MA., Rinde-Hoffman, D., Wigger, M., Wang, YS., Wolf, T., Arnold, PJ., Sninsky, J., Berman, P. Routine Surveillance of Heart Transplant Recipients with Gene Expression Profiling: Lack of an Impact of Race on Outcomes. 2017 American Transplant Congress. April 29-May 3, 2017; Chicago, IL. Poster
- [Result] Shah, P. et al: Outcomes with Gene Expression Profiling for Cardiac Transplant Recipients Within North America. 2016 ISHLT 36th Annual Meeting and Scientific Sessions. April 27-30, 2016; Washington, DC.
- [Result] Uriel, N. et al; Utility of Gene Expression (AlloMap Score) in Antibody Mediated Rejection Detection. 2016 ISHLT 36th Annual Meeting and Scientific Sessions. April 27-30, 2016; Washington, DC.